CLINICAL TRIAL: NCT04642469
Title: A Phase III, Randomized, Multicenter, Double-blind, Placebo-controlled Study of Durvalumab for the Treatment of Stage II-III NSCLC Patients With Minimal Residual Disease Following Surgery and Curative Intent Therapy.
Brief Title: Phase III Study to Determine Efficacy of Durvalumab in Stage II-III Non-small Cell Lung Cancer (NSCLC) After Curative Intent Therapy.
Acronym: MERMAID-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D910MC00001; 2020-000612-30 (EudraCT Number)
Record Dates: First submitted 2020-11-03; First posted 2020-11-24 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Non- Small Cell Lung
Keywords: NCSLC; Double-blind; PD-L1; MEDI4736; Durvalumab; DFS; OS; MRD+; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind and open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): Intravenous administration of Durvalumab
  Interventions: Drug: Durvalumab
- Placebo (Placebo Comparator): Intravenous administration of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Durvalumab — Intravenous administration of Durvalumab
  Other Names: Medi4736
  Arms: Durvalumab
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This is a Phase III double-blind, placebo-controlled study of Durvalumab versus Placebo in patients with stage II-III NSCLC who are MRD-positive following curative intent therapy.

DETAILED DESCRIPTION:
This is a Phase III, randomized, multicenter, double-blind, placebo-controlled, study to evaluate the efficacy and safety of durvalumab adjuvant therapy compared to placebo in patients with completely resected stage II-III NSCLC who have undergone curative intent therapy (complete resection ± neoadjuvant and/or adjuvant therapy), who have no evidence of Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1-defined disease recurrence, and who become MRD+ during surveillance period.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICFs and in the protocol.
2. Provision of signed and dated, written informed consent form prior to any mandatory study-specific procedures, sampling, and analyses.
3. Provision of signed and dated written optional genetic informed consent prior to collection of the optional sample for genetic analysis. This consent should be signed at the time of second screening. This optional sample and analyses are separate from the mandatory genetic testing consent included in ICF1.

   The following criteria must have been met at the time of surgery or at the time of the curative intent therapy (first screening):
4. Age ≥18 years at the time of screening (ICF1);
5. Male and/or female
6. Histologically confirmed NSCLC with resectable stage II-III disease who have undergone curative intent therapy (complete resection of the primary tumor ± neoadjuvant and/or adjuvant therapy) per SoC.

   Select stage IIIB (ie, T3N2 or T4N2) patients will be eligible, provided they are upstaged to T3N2 or T4N2 based on confirmed pathology after surgery. Patients who are staged as T3N2 or T4N2 prior to surgery are not eligible.
7. A contrast-enhanced CT/MRI scan of the chest and abdomen (including liver and adrenal glands) along with brain MRI (preferred) or brain CT with IV contrast must have been done for surgical planning prior to surgery. It is recommended that patients undergo combined FDG-PET (18F-Fluoro-deoxyglucose positron emission tomography) and CT scan (computerized tomography) within the 6 weeks prior to surgery in order to rule out detectable extrathoracic, extracranial metastasis and to assess for potential mediastinal lymph node involvement prior to surgery. If the positron emission tomography (PET) scan was not performed, or data from a PET is not available, patients may still be enrolled into the study provided appropriate imaging (CT/MRI) is performed prior to randomization.
8. Complete resection of the primary NSCLC is mandatory. Invasive (pre-operative or intra-operative) exploration of hilar and mediastinal lymph nodes must have been performed to confirm primary tumor nodal status (prior to or after surgery). Surgical resection of the primary NSCLC can occur by open thoracotomy or by video-assisted thoracic surgery (VATs) and resection can be achieved by segmentectomy, lobectomy, sleeve resection, bilobectomy or pneumonectomy. Patients undergoing wedge resection are not eligible for this study.

   Criteria for prior systemic chemotherapy/radiotherapy:
9. Patients should have completed (or be undergoing) curative intent therapy (surgery ± neoadjuvant and/or adjuvant therapy; adjuvant therapy can include PORT) with exceptions noted below:

   Patients who discontinue chemotherapy and/or PORT for toxicity prior to completion of all planned therapy are eligible.

   Patients who have not received any neoadjuvant and/or adjuvant chemotherapy, and meet all other eligibility criteria, may be eligible under the following circumstances:
   * All patients who are eligible for adjuvant chemotherapy MUST be offered adjuvant chemotherapy.
   * The patient has declined adjuvant chemotherapy, and in the opinion of the Investigator, this is the patient's final decision after receiving appropriate information and adequate time to make the decision. The patient's refusal of adjuvant chemotherapy must be documented.
   * If in the view of the Investigator, adjuvant chemotherapy is contraindicated due to an underlying intercurrent illness/laboratory abnormality, which is not considered reversible within a reasonable timeframe for the patient to be eligible for adjuvant therapy, which must be documented.

   Criteria assessed prior to and at the start of surveillance:
10. Confirmation of suitable biosamples for WES and central PD-L1 testing. Resected tumor tissue and whole blood samples must be provided to the diagnostic laboratory for WES of tumor and germline DNA, respectively as soon as possible following pathology confirmation. Samples must be sent no later than 1-2 weeks after completion of adjuvant therapy or 3-5 weeks after surgery (if no adjuvant therapy is given) for development of the Sponsor-approved personalized panel for MRD detection at a central reference laboratory. Germline sequencing of whole blood is mandatory. Resected tumor tissue must also be provided for PD-L1 testing at a central reference laboratory (see inclusion criteria 15).
11. Post-adjuvant therapy or post-surgery (if no adjuvant therapy is given) CT scan of the chest and abdomen (including liver and adrenal glands) and brain MRI [preferred] or brain CT with IV contrast should be available to confirm no evidence of metastasis. If scans were not performed post-curative intent therapy, additional scans must be done prior to start of surveillance.
12. Consents to be accessible for q6w±3d plasma sample collection for MRD evaluation and for q12w±1w CT scans during the 96-week surveillance period.
13. The plasma sample that marks the start of surveillance must be collected 8±1 weeks after completion of adjuvant therapy (if administered) or 12±1 weeks after surgery (where adjuvant therapy is not given).

    * A patient who is determined to be MRD- based on analysis of this plasma sample (ie, MRD- at the start of surveillance) may continue in surveillance provided all other eligibility criteria are met.
    * A patient who is determined to be MRD+ based on analysis of this plasma sample (ie, MRD+ at the start of surveillance) may be eligible for immediate randomization provided all other eligibility criteria are met.

    A patient who becomes MRD+ during surveillance is eligible to enter the second screening period and may be randomized in the study if all other eligibility criteria are met.

    Criteria for second screening prior to randomization to treatment:
14. CT scan of the chest and abdomen (including liver and adrenal glands) and brain MRI [preferred] or brain CT with IV contrast performed within the 28 days ± 7 days prior to randomization to confirm no evidence of RECIST 1.1-defined disease recurrence and/or metastasis.
15. Known tumor PD-L1 status determined at a central reference laboratory testing service using a validated Ventana SP263 PD-L1 immunohistochemistry (IHC) assay prior randomization. Patients with unknown PD-L1 status are not eligible for the study.
16. WHO/Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
17. Complete post-operative wound healing must have occurred prior to randomization; patients must have recovered from all acute, reversible toxic effects from prior treatments (excluding alopecia) that could potentially adversely impact further administration of durvalumab/placebo according to the Investigator's judgment.
18. Must have recovered from all acute, reversible toxic effects from chemotherapy that could potentially adversely impact further administration of durvalumab or placebo according to the Investigator's judgment
19. Adequate organ and marrow function as described in the protocol.
20. Must have a life expectancy of at least 12 weeks Weight
21. Body weight >30 kg Inclusion criteria assessed prior to entering the observation period
22. No evidence of RECIST 1.1-defined disease recurrence or metastasis confirmed by CT scan of the chest and abdomen (including liver and adrenal glands) and a brain MRI (preferred) or brain CT with IV contrast.
23. MRD- status, as determined by testing the last plasma sample collected during the 96-week surveillance period.

Exclusion Criteria:

Diagnostics assessments:

1. EGFR and/or ALK mutant as assessed either from the tumor biopsy taken prior to surgery or the resected tumor tissue. Testing must be performed using a wellvalidated, local regulatory-approved test. EGFR/ALK may be tested centrally if local testing is unavailable.
2. Mixed small cell and NSCLC histology.
3. Require re-resection or are deemed to have unresectable NSCLC by amultidisciplinary evaluation that must include a thoracic surgeon who performs lung cancer surgery as a significant part of their practice.
4. Baseline imaging demonstrating unequivocal evidence of RECIST 1.1-defined disease recurrence or evidence of clinical recurrence outside of imaging prior to randomization. In the event of lymphadenopathy on imaging that would lead to exclusion, histopathological confirmation of lymph node metastasis should be obtained prior to excluding a patient from the study. If pathological confirmation of lymph node metastasis is not technically feasible and imaging appearance are deemed unequivocal for relapse, the patient will be excluded.

   Medical conditions
5. History of allogeneic organ or bone marrow transplantation.
6. Non-leukocyte-depleted whole blood transfusion in 120 days of genetic sample collection
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or

   Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   Patients with vitiligo or alopecia Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement Any chronic skin condition that does not require systemic therapy Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician Patients with celiac disease controlled by diet alone
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active ILD, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
9. History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in-situ without evidence of disease
10. History of active primary immunodeficiency
11. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B virus (HBV) (known positive HBV surface antigen (HBsAg) result), hepatitis C virus (HCV), or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
12. Known allergy or hypersensitivity to any of the IPs or any of the IP excipients Prior/concomitant therapy
13. Received any IO therapy in the adjuvant setting or any prior exposure to durvalumab.
14. Received any radiotherapy in the neoadjuvant setting.
15. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
16. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of IP.
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
18. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of IP. The following are exceptions to this criterion:

    Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) Prior/concurrent clinical study experience
20. Previous IP assignment in the present study
21. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
22. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

    Other exclusions
23. Female patients who are pregnant or breastfeeding.

    - Female patients who become pregnant during the study will be withdrawn from surveillance and are not eligible for randomization.
24. Male or female patients of reproductive potential who are not willing to employ effective birth control at the time of entry into second screening (initiated with the signing of ICF2a) until 90 days after the last dose of IP (See Appendix H).
25. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, Principal Investigator — SCRI Development Innovations, LLC; Charles Swanton, Principal Investigator — Francis Crick Institute
Locations (102):
- United States (10):
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Daytona Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Punta Gorda, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, Minneapolis, Minnesota
  - Research Site, Spartanburg, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
- Research Site, Buenos Aires, Argentina
- Australia (3):
  - Research Site, Camperdown
  - Research Site, Melbourne
  - Research Site, St Leonards
- Belgium (2):
  - Research Site, Hasselt
  - Research Site, Roeselare
- Brazil (5):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, Vitória
- Canada (5):
  - Research Site, Victoria, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, Kingston, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- France (4):
  - Research Site, Marseille
  - Research Site, Pessac
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
- Greece (5):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Holargos, Athens
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Jordan
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Törökbálint
- India (2):
  - Research Site, Bengaluru
  - Research Site, New Delhi
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (6):
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (9):
  - Research Site, Bunkyō City
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Maastricht
  - Research Site, Zwolle
- Research Site, Lima, Peru
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Santiago de Compostela
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Malatya
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910MC00001&attachmentIdentifier=87ff8c14-5d81-4b1e-917e-b062d63d134e&fileName=d910mc00001-csp-v2_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910MC00001&attachmentIdentifier=1109be20-4d3e-4900-8faa-73cd619fda9e&fileName=d910mc00001-sap-ed-2_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910MC00001&attachmentIdentifier=2ca4ff82-8586-4b4b-b79e-ca8e45144b18&fileName=d910mc00001-abbreviated-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III multicenter, double-blind, placebo-controlled study was conducted in participants with Stage II to III non-small cell lung cancer (NSCLC) at 21 sites in 13 countries (Australia, Brazil, Czech Republic, France, Greece, Hungary, Israel, Italy, Japan, Spain, Taiwan, Turkey, and United States). First participant was enrolled on 30-Nov-2020 and final data cut-off (DCO) date was 31 May 2023.
Pre-assignment Details: 30 participants were randomized in a 1:1 ratio to receive durvalumab monotherapy or placebo in the study.
Groups:
- Durvalumab: Participants received durvalumab 1500 milligram (mg) via intravenous (IV) infusion over 60 minutes, once every 4 weeks (q4w) for a maximum of 26 cycles, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Placebo: Participants received matching placebo via IV infusion over 60 minutes, once q4w for a maximum of 26 cycles, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Durvalumab | Placebo
Started | 15 | 15
Completed | 0 | 1
Not Completed | 15 | 14
Not completed — Failure to meet inclusion/exclusion criteria | 1 | 0
Not completed — Death | 1 | 2
Not completed — Study/site closed following amendment 1 | 11 | 11
Not completed — Other | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (8.6) | 66.7 (10.3) | 63.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 5 | 8
  White | 7 | 7 | 14
  Other | 1 | 0 | 1
  Missing | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: DFS was defined as the time from the date of randomization until any one of the following events, whichever occurred first: Date of disease recurrence using Investigator assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 OR Date of death from any cause.
Time Frame: Every 8 weeks (q8w) ± 1 week until Week 48, then every 12 weeks (q12w) ± 1 week until appearance of RECIST 1.1-defined disease recurrence or follow-up, up to 16.6 months
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 15 | 15
Months | 3.9 [3.515 to NA] — NA indicates that upper limit of confidence interval was not estimable due to insufficient number of participants with events at study closure and due to limited duration of follow-up. | 2.0 [1.643 to 3.910]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event was any untoward medical occurrence (other than progression of the malignancy under evaluation) in a participant or clinical study participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An SAE was an AE that occurred during any study phase and fulfilled one or more of the following criteria: Resulted in death, was immediately life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital abnormality or birth defect, was an important medical event that might jeopardize the participant or might require medical treatment to prevent one of the outcomes listed above, AEs for malignant tumors reported during a study, malignant tumors that - as part of normal, if rare, progression - underwent transformation.
Time Frame: From start of study treatment (Day 1) up to 90 days after last dose of study treatment, approximately 21.4 months
Population: The Safety Analysis Set included all randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 14 | 15
Participants
  Any AEs | 13 | 10
  Any SAEs | 1 | 1

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse events (TEAEs) were collected from start of study treatment (Day 1) up to 90 days after last dose of study treatment, approximately 21.4 months. All-cause mortality was collected from start of randomization (Day 0) up to completion of study, approximately 30 months.
Description: The Safety Analysis Set included all randomized participants who received any amount of study treatment. All-cause mortality was reported in FAS.
Arm/Group | Durvalumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/15 | 2/15
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/15
Other Adverse Events (participants affected / at risk) | 13/14 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=14) | Placebo (N=15)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=14) | Placebo (N=15)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Tachyphrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor closed enrollment to the study early due to treatment landscape changes. Interpretation of study outcomes were limited by the resulting small sample size and limited duration of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04642469/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT04642469/SAP_001.pdf